CLINICAL TRIAL: NCT03944083
Title: Emotional Dysregulation in Children With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Children With ADHD and Emotional Dysregulation
Acronym: MOODY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Lovisenberg Diakonale Hospital (Other)
Responsible Party: Principal Investigator, Pål Zeiner, Project manager, Oslo University Hospital
Other Study IDs: 2017/135
Record Dates: First submitted 2019-05-06; First posted 2019-05-09 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Attention Deficit Hyperactivity Disorder; Disruptive Mood Dysregulation Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Hair samples analyzed on cortisol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ADHD with and without DMDD: ADHD with DMDD versus ADHD without DMDD. Observational study at referral and after 6 and 12 months.
  Interventions: Other: Treatment as usual for ADHD

INTERVENTIONS:
Other: Treatment as usual for ADHD — Children are given treatment according to diagnostic conclusion and clinical recommendations.

SUMMARY:
Studies have shown that children with Attention Deficit Hyperactivity Disorder (ADHD) and emotional dysregulation are characterized by high severity of ADHD, comorbid behavior disorders and increased risk of chronic difficulties.

New studies have shown promising results by focusing on improving emotional regulation. We lack knowledge about differences in symptom patterns, stability of symptoms over time, comorbid disorders, neurocognitive functions, knowledge and regulation of emotions, psychosocial risk factors and reactions to stress.

Children 6 to 12 years admitted to specialist and diagnosed with ADHD will be recruited. ADHD children with and without emotional dysregulation defined as fullfilling the criteria for the diagnosis Disruptive Mood Dysregulation Disorder (DMDD) with regard to differences in symptom patterns, stability of symptoms over time, comorbid disorders, neurocognitive functions, knowledge and regulation of emotions, psychosocial risk factors and reactions to stress..

DETAILED DESCRIPTION:
Children referred to outpatient psychiatric service will be informed about the study and asked to participate. The clinical assessments in the study will be those that are recommended as good clinical practice, so results will be included in the diagnostic work for the patient.

The data security will follow the Norwegian rules and be monitored by REC and the Data Inspectorate of the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Referred to outpatient psychiatric service.
* IQ within normal range.
* Child and parents: Good enough understanding of Norwegian language to give valid answers in interviews and tests.

Exclusion Criteria:

* IQ below normal range.
* Child and parents: Not good enough understanding of Norwegian language to give valid answers in interviews and tests.
* Unresolved crisis in the family.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children referred to outpatient psychiatric service
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Attention Deficit Hyperactivity Disorder-Rating Scale total score | 12 months
  Symptom score. Measure difference from baseline. Lower score means improvement.
Disruptive Mood Dysregulation Disorder total symptom questionnaire score | 12 months
  Symptom score. Symptom score. Measure difference from baseline. Lower score means improvement.
Number of other comorbid disorders in psychiatric interview | Baseline
  DSM-5 diagnoses: Types and number of diagnoses. More diagnoses means more complex disorder.
Affect recognition total score | Baseline
  Test from NEPSY II. Comparison With norms. Difference from norm reported.
Hair cortisol Level | Baseline
  Cortisol level over time

CONTACTS AND LOCATIONS:
Overall Officials: Pål Zeiner, PhD, Principal Investigator — Head of child psychiatric research
Locations (1):
- Nic Waal's Institute, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
The data are on patients. We need to decide whether or not anonymous data can be shared with other researchers.